CLINICAL TRIAL: NCT01804400
Title: A Randomized, Double-blind, Placebo-controlled Three-period Incomplete Cross Over Study to Compare the Efficacy of QAW039 Alone and in Combination With Montelukast in Patients With Allergic Rhinitis Using an Environmental Exposure Chamber
Brief Title: A Clinical Trial to Test How Well Two Drugs, QAW039 and Montelukast Work Both Individually and Together, to Target Allergic Rhinitis Using an Environmental Exposure Chamber
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CQAW039A2212; 2012-001389-14 (EudraCT Number)
Record Dates: First submitted 2012-10-04; First posted 2013-03-05 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — fevipiprant; montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- QAW039 + Montelukast (Experimental)
  Interventions: Drug: QAW039; Drug: Montelukast; Drug: Placebo
- QAW039 Once a day (q.d.) (Experimental)
  Interventions: Drug: QAW039; Drug: Placebo
- QAW039 Twice a day (b.i.d.) (Experimental)
  Interventions: Drug: QAW039; Drug: Placebo
- Montelukast (Active Comparator)
  Interventions: Drug: Montelukast; Drug: Placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: QAW039
  Arms: QAW039 + Montelukast; QAW039 Once a day (q.d.); QAW039 Twice a day (b.i.d.)
Drug: Montelukast
  Arms: Montelukast; QAW039 + Montelukast
Drug: Placebo

SUMMARY:
This study will assess the safety and efficacy of QAW039 alone and in combination with Montelukast in patients with allergic rhinitis (hay fever) using an environmental exposure chamber.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-65 years inclusive, with a clinical history of intermittent allergic rhinitis with seasonal onset and offset of nasal allergy symptoms during each of the last two grass pollen allergy seasons.
* A positive skin prick test at Visit 1 to dactylis glomerata with a wheal diameter equal to or greater than 3 mm and a negative control with a wheal diameter of zero. A positive skin prick test within 12 months prior to Visit 1 is also acceptable.
* FEV1 measured by spirometry must be ≥80% of their predicted value at screening. If the patient does not achieve ≥80% of their predicted value this may be repeated prior to the EEC challenge at visit 2.
* TNSS score ≥6 on at least one assessment during the 2h EEC challenge at Screening.

Exclusion Criteria:

* Use of other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer; or longer if required by local regulations, and for any other limitation of participation in an investigational trial based on local regulations.
* Pregnant or nursing (lactating) women,
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using effective methods of contraception during dosing of study treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2012-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change in Total Nasal Symptom Score from baseline at 14 days | Baseline, Day 14
  Total Nasal Symptom Score (TNSS) averaged over the last two hours (2-4h) of exposure following 14 days treatment with QAW039 and/or Montelukast or matched placebo

SECONDARY OUTCOMES:
Change in Total Ocular Symptom score from Baseline at 14 days | Baseline, Day 14
  Total Ocular Symptom Score (TOSS), defined as the sum of ocular symptoms of eye tearing, itching, watery eyes and redness, each of which is scored on a scale from 0 and 3
Change in Nasal Flow from baseline at 14 days | Prior to, and every 60 min during allergen exposure period
  Measured using rhinomanometry Flow rates at 150 Pa will be obtained separately for the right and left nostrils (cm^3/second). The sum of the flow rates of both nostrils will be calculated from the two measurements
Change in Nasal excretion weight from baseline at 14 days | Baseline, Day 14
  Total weight of tissues (before and after use)
Change in Forced Expiratory Volume in 1 Second (FEV1) from baseline at 14 days | Baseline, Day 14
  Change in FEV1 from Baseline
Change in Forced Vital Capacity (FVC) from baseline at 14 days | Baseline, Day 14
  Change in FVC from Baseline
Change in FEV1/FVC at from baseline at 14 days | Baseline, Day 14
  Change in FEV1/FVC from Baseline
Plasma Concentration maximum (Cmax) | Day 1-14
  Determined at steady state in plasma
Plasma Concentration Minimum (Cmin) | Day 1-14
  Determined at steady state in plasma
Plasma Concentration Average (Cav) | Day 1-14
  Determined at steady state in plasma
Time of Cmax (Tmax) | Day 1-14
  Determined at steady state in plasma
Area Under Curve (AUCtau) | Day 1-14
  Determined at steady state in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Hanover, Germany